CLINICAL TRIAL: NCT05840627
Title: The Effect of Daily Consumption of a Fruit Juice on Acute Satiety Response and Gut Microbiota Changes in Healthy Adults
Brief Title: Acute Satiety and Metabolic Response of Daily Consumption of a Fruit Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: cLabel+
Record Dates: First submitted 2023-03-06; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Healthy
MeSH Terms: interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruit juice (Experimental)
  Interventions: Other: Fruit juice

INTERVENTIONS:
Other: Fruit juice — Daily consumption of 200 mL of fruit juice at lunch for 14 consecutive days, provided by the research team.

SUMMARY:
The "cLabel+ Innovative natural, nutritious and consumer-oriented clean label food" is a research and technological development project centered on responding to the challenges facing the food industry. It is focused on the concept of "clean label", which emerges as one of the major current trends in the sector, given the growing number of consumers who are increasingly aware and eager for information, who are looking for alternative, more transparent and natural food products.

Thus, one of the aims of the cLabel+ project is to research the macronutrients and phenolic compounds present in food matrices and achieve a clean label positioning for the final products developed. This single group assignment clinical trial aims to evaluate the effect of daily consumption of a fruit juice, developed as part of the collaborative project cLabel+, on gut microbiota composition and diversity in healthy adults. It is also intended to study the acute metabolic effect, namely in terms of appetite control, and lipid and glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Adults (age ≥ 18 years)
* Filling informed consent

Exclusion Criteria:

* Obesity (body mass index ≥ 30.0 kg/m2).
* Daily consumption of fruit juices in the month prior to the start of the study.
* Individuals with diagnosed food allergies or intolerances to the components being tested.
* Use of pro/prebiotics or fibre as a dietary supplement or any food/molecule that modifies intestinal transit time 6 weeks before recruitment.
* Use of laxatives 6 weeks before recruitment.
* Recent weight loss or weight gain of more than 10% in the last 3 months.
* Adherence to restrictive weight loss diets or specific dietary pattern (e.g., palaeolithic diet, Atkins, flexitarian, ketogenic, vegan).
* Diagnosis of gastrointestinal pathology, hormonal or thyroid pathology, autoimmune diseases, chronic use of corticosteroids, psychiatric disease, or diabetes mellitus.
* Having taken antibiotics within the 12 weeks prior to beginning the study.
* Excessive consumption of alcoholic beverages (>14 and >8 units/week for men and women, respectively).
* Pregnant or breastfeeding.
* Participation in another clinical trial within the past 3 months that the Principal Investigator believes may compromise the results of the trial (e.g., clinical trial with an effect on the composition and diversity of the gut microbiota).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota characterization | 14 days
  Differences in gut microbiota taxonomic characterization from baseline to the end of the intervention.
Changes in gut microbiota diversity | 14 days
  Difference in gut microbiota Shannon index, from baseline to the end of intervention.
Changes in the iAUC (pmol/L*min) for ghrelin | 14 days
  Ghrelin will be measured in fasting and every 30 minutes up to 3 hours. The iAUC (pmol/L*min) for ghrelin will be calculated based on the concentration curve following consumption of the fruit juice.
Changes in the iAUC (pmol/L*min) for glucagon-like peptide-1 (GLP-1) | 14 days
  GLP-1 will be measured in fasting and every 30 minutes up to 3 hours. The iAUC (pmol/L*min) for GLP-1 will be calculated based on the concentration curve following consumption of the fruit juice.
Changes in the iAUC (pmol/L*min) for peptide YY (PYY) | 14 days
  PYY will be measured in fasting and every 30 minutes up to 3 hours. The iAUC (pmol/L*min) for PYY will be calculated based on the concentration curve following consumption of the fruit juice.

SECONDARY OUTCOMES:
Changes in fasting glucose | 14 days
  Changes in fasting glucose, measured in mg/dL, from baseline to the end of intervention.
Changes in fasting insulin | 14 days
  Changes in fasting insulin, measured in mg/dL, from baseline to the end of intervention.
Changes in HOMA-IR | 14 days
  Changes in HOMA-IR from baseline to the end of intervention.
Changes in total cholesterol | 14 days
  Changes in total cholesterol, measured in mg/dL, from baseline to the end of intervention.
Changes in LDL cholesterol | 14 days
  Changes in LDL cholesterol, measured in mg/dL, from baseline to the end of intervention.
Changes in HDL cholesterol | 14 days
  Changes in HDL cholesterol, measured in mg/dL, from baseline to the end of intervention.
Changes in triacylglycerols | 14 days
  Changes in triacylglycerols, measured in mg/dL, from baseline to the end of intervention.
Changes in high sensitivity PCR | 14 days
  Changes in high sensitivity PCR, measured in mg/dL, from baseline to the end of intervention.
Changes in expired breath H2 | 14 days
  Changes in expired breath H2, measured in ppm, from baseline to the end of intervention.
Changes in expired breath CH4 | 14 days
  Changes in expired breath CH4, measured in ppm, from baseline to the end of intervention.
Changes in faecal butyrate | 14 days
  Changes in faecal butyrate, measured in M, from baseline to the end of intervention.
Changes in faecal acetate | 14 days
  Changes in faecal acetate, measured in M, from baseline to the end of intervention.
Changes in faecal alkaline phosphatase (ALP) | 14 days
  Changes in faecal ALP, measured in mg/g faeces, from baseline to the end of intervention.
Changes in faecal LPS | 14 days
  Changes in faecal LPS, measured in EU/mL, from baseline to the end of intervention.
Changes in faecal calprotectin | 14 days
  Changes in faecal calprotectin, measured in µg/g faeces, from baseline to the end of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- NOVA Medical School|Faculdade de Ciências Médicas, Universidade NOVA de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No